CLINICAL TRIAL: NCT02776761
Title: Hantaan Virus Plasmid DNA Vaccine (Expressing Gn and Gc Antigens; E. Coli) [HTNV Vaccine] and Puumala Virus Plasmid DNA Vaccine (Expressing Gn and Gc Antigens; E. Coli; Ajinomoto Bio-Pharma Services) [PUUV Vaccine] Administered Via Stratus Needle-free Injection System (PharmaJet, Inc.)
Brief Title: A Single-blind Study to Evaluate the Safety, Tolerability, and Immunogenicity of a Hantaan Puumala Virus DNA Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: S-15-40; WRAIR 2289 (Other: WRAIR)
Record Dates: First submitted 2016-05-13; First posted 2016-05-18 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Hantaan Virus

STUDY DESIGN:
Intervention Model Description: Study will enroll 3 randomized groups of 9 subjects for a total of 27 subjects. Every subject will receive a total of 3 vaccinations. Subjects will be blinded to the group they are randomized to. Each vaccination consists of 2 administrations of 1 mg (left/right deltoid) for a total of 2 mg/vaccination. Group 1 will be vaccinated with the HTNV vaccine, pWRG/HTN-M (co). Group 2 will be vaccinated with the PUUV vaccine, pWRG/PUU-M (s2). Group 3 will be vaccinated with a combined HTNV/PUUV vaccines. Each group will be vaccinated on Days 0, 28, and 56. An optional 4th vaccination on Day 168 with follow-up on Day 196. All doses will be administered with PharmaJet Stratis device. All subjects to be followed until at least 3 months post last vaccination with Day 252 the final study visit (a 12-month, optional follow-up visit may be requested approximately on Day 365). Subjects will complete postinjection memory aids for 7 days after each vaccination.
Who Masked: Participant
Masking Description: Subjects will be blinded to the vaccine(s) they are receiving. All subjects will receive active product; there is no placebo control group.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hantaan Vaccine: (Experimental): 1 mg in 0.5 mL per administration, 2 administrations per vaccination, total injected volume 1 mL per vaccination (for 2.0 mg dose)
  Interventions: Biological: Hantaan Vaccine:
- Puumala Vaccine: (Experimental): 1 mg in 0.5 mL per administration, 2 administrations per vaccination, total injected volume 1 mL per vaccination (for 2.0 mg dose)
  Interventions: Biological: Puumala Vaccine
- Hantaan/Puumala Vaccine (Experimental): The HTNV and PUUV vaccine will be combined (equal volumes) before use: 1 mg in 0.5 mL per administration, 2 administrations per vaccination, total injected volume 1 mL per vaccination (for 2.0 mg dose)
  Interventions: Biological: Hantaan/Puumala Vaccine

INTERVENTIONS:
Biological: Hantaan Vaccine: — DNA Vaccine 2.0 mg/1 mL phosphate-buffered saline
  Arms: Hantaan Vaccine:
Biological: Puumala Vaccine — DNA Vaccine 2.0 mg/1 mL phosphate-buffered saline
  Arms: Puumala Vaccine:
Biological: Hantaan/Puumala Vaccine — DNA Vaccine 2.0 mg/1 mL phosphate-buffered saline
  Arms: Hantaan/Puumala Vaccine

SUMMARY:
This is a single-center, randomized, single-blinded study of the Hantaan virus HTNV DNA vaccine alone, Puumala virus PUUV DNA vaccine alone, and mixed Hantaan/Puumala HTNV/PUUV DNA vaccines delivered intramuscularly IM by the needle-free PharmaJet Stratus DSJI device.

DETAILED DESCRIPTION:
Investigational HTNV and PUUV DNA vaccines, manufactured in accordance with cGMP guidelines by Ajinomoto Bio-Pharma Services (California), from their respective drug substances, pWRG/HTN-M(co) and pWRG/PUU-M(s2),were constructed on a well-characterized plasmid backbone, pWRG7077. These plasmid DNA vaccines will be delivered IM using the needle-free, disposable syringe jet injection device (PharmaJet Stratis). Subjects will be randomized into 3 groups of 9 subjects each for a total of 27 subjects. Each subject will receive a total of 3 vaccinations. Group 1 vaccine will consist of 2 administrations of 1 mg of HTN plasmid (left and right deltoid) for a total of 2 mg/vaccination. Group 2 vaccine will consist of 2 administrations of 1 mg of PUU plasmid (left, right deltoid) for a total of 2 mg/vaccination. Group 3 vaccine will consist of a 1:1 mixture of HTNM and PUU vaccines (left, right deltoid) for a total of 2 mg/vaccination (1 mg/vaccination of each DNA). Vaccinations will be administered on Days 0, 28, and 56. There will be an optional 4th vaccination on Day 168 dependent on subject availability for the additional follow-up visit on Day 196, tolerability of the vaccinations to date, and investigator discretion. Volunteers will be invited back for the 4th vaccination to determine if a booster dose results in increased immunogenicity and seroconversion. All subjects will be followed until Day 252 (9 months). A Day 365 follow-up visit, for an immunogenicity draw only, may be requested dependent on immunogenicity results shortly after this final date, generally within 4 weeks of the Day 252 visit or once the assays can be completed. Subjects may be allowed to receive other licensed vaccinations or enroll in other clinical trials after the Day 252 visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or nonpregnant, nonlactating female, ages 18-49 (inclusive) at the time of screening
* Have provided written informed consent before screening
* Free of clinically significant health problems as determined by pertinent medical history and clinical examination prior to entry into the study
* Available and able to participate for all study visits and procedures
* Females, if not abstinent, are known to be at least 1 year post-menopausal (defined as no menses for 12 consecutive months) or willing to use an effective method of contraception (eg, hormonal contraception to include oral and implantable options, diaphragm, cervical cap, intrauterine device, condom, or anatomical sterility [self or partner]) for the duration of study participation (from the date of screening) until at least 3 months after the last injection
* Negative hantavirus PsVNA test result at screening

Exclusion Criteria:

* History or serologic evidence of prior infection with any hantavirus or prior participation in an HTNV or PUUV vaccine trial
* History of severe local or systemic reactions to any vaccination or a history of severe allergic reactions
* Ongoing participation in another clinical trial (subjects continuing through Day 365 will not join other new studies until their final visit)
* Receipt of licensed vaccines within 14 days before or after immunization (30 days for live vaccines)
* Ability to observe possible local reactions at the eligible injections sites (deltoid region) is, in the opinion of the investigator, unacceptably obscured due to a physical condition or permanent body art
* Acute or chronic, clinically significant hematologic, pulmonary, cardiovascular, or hepatic or renal functional abnormality as determined by the investigator based on medical history, physical exam, and/or laboratory screening test
* Pregnant or lactating female, or female who intends to become pregnant during the study period
* Administration of immunoglobulins and/or any blood products within the 120 days preceding study entry or planned administration during the study period Blood donation for human use (eg, American Red Cross or other similar blood drives) within the 56 days preceding study entry or planned administration during the study period
* Any confirmed evidence of hepatitis B or C infection
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection
* Administration of chronic (defined as more than 14 days) immunosuppressants or other immune-modifying drugs within 6 months of study entry
* For corticosteroids, this will mean prednisone, or equivalent, greater than or equal to 0.5 mg/kg/day
* Intranasal, inhaled, and topical steroids are allowed (daily inhaled steroids for treatment of asthma are NOT allowed)
* Any chronic or active neurologic disorder, including seizures and epilepsy, excluding a single febrile seizure as a child
* Suspected or known current alcohol and/or illicit drug abuse
* Unwilling to allow storage and use of blood for future hantavirus-related research
* Any other significant finding that in the opinion of the investigator would increase the risk of the individual having an adverse outcome from participating in this study

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2016-08-30 (Actual); Primary Completion 2017-09-27 (Actual); Study Completion 2017-09-27 (Actual)

PRIMARY OUTCOMES:
Hantaan Vaccine: Number of Adverse Events | 365 days
  Number of adverse events.
Puumala Vaccine: Number of Adverse Events | 365 days
  Number of adverse events.
Hantaan/Puumala Vaccine: Number of Adverse Events | 365 days
  Number of adverse events.

SECONDARY OUTCOMES:
Hantaan Vaccine (50) immunogenicity | 365 days
  Pseudovirion neutralization assay 50% titer
Puumala Vaccine (50) immunogenicity | 365 days
  Pseudovirion neutralization assay 50% titer
Hantaan/Puumala Vaccin (50) immunogenicity | 365 days
  Pseudovirion neutralization assay 50% titer
Hantaan Vaccine (80) immunogenicity | 365 days
  Pseudovirion neutralization assay 80% titer
Puumala Vaccine (80) immunogenicity | 365 days
  Pseudovirion neutralization assay 80% titer
Hantaan/Puumala Vaccin (80) immunogenicity | 365 days
  Pseudovirion neutralization assay 80% titer
Hantaan Vaccine (80) immunogenicity | 84 days
  Plaque-reduction neutralization test (PRNT) comparing Day 0 to Day 84
Puumala Vaccine (80) immunogenicity | 84 days
  Plaque-reduction neutralization test (PRNT) comparing Day 0 to Day 84
Hantaan/Puumala Vaccin (80) immunogenicity | 84 days
  Plaque-reduction neutralization test (PRNT) comparing Day 0 to Day 84

CONTACTS AND LOCATIONS:
Overall Officials: Kristopher Paolino, MD, Principal Investigator — Walter Reed Army Institute of Research (WRAIR)
Locations (1):
- WRAIR Clinical Trials Center, Silver Spring, Maryland, United States